CLINICAL TRIAL: NCT06677242
Title: Serous Endometrial Intraepithelial Carcinoma (SEIC): Prospective Registration Study
Acronym: SEIC
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ciska Slaager, MD, PhD student and resident in gynaecology, Erasmus Medical Center
Other Study IDs: OZBS82.24252
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Serous Endometrial Intraepithalial Carcinoma; SEIC
Keywords: Sereus endometrial intraepithelial carcinoma; SEIC; Endometrial cancer; Premalignant neoplasms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Blood Specimen Collection; Vaginal Smears

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood serum for circulating tumor DNA and additional PAP-smear for genome-wide methylation sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Blood sample (serum) for circulating tumor DNA and cervical smear for genome-wide methylation sequencing — These are additional tests, added to the observational study to collect information on tumor characteristics and to pursue early detection of this diagnosis.

SUMMARY:
Background: Serous endometrial intra-epithelial carcinoma (SEIC) is a rare condition affecting the lining of the uterus. It's a pre-cancerous change that might lead to cancer if not treated. Doctors aren't sure of the best way to manage it because it's so uncommon. A previous study looked at past cases in the Netherlands from 2012 to 2020. This study found that none of the 23 women with SEIC had their cancer spread during surgery, and none had a recurrence in the following three years. This suggests that a simpler surgery might be safe for patients with SEIC.

Methods: Information on disease details from patients who agree to participate in our study will be collected. All participants will fill out online forms and health questionnaires at several points: when they join the study, and again at six months, two years, and five years after their diagnosis. During the years after diagnosis, various details like health status, test results, treatments will be checked in the electronic medical record.

Results: This study is just starting, with the first patients expected to join on January 1, 2025.

Conclusion: A large international study is created to track SEIC patients over time. This will help us learn more about the condition and improve treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Serous endometrial intra-epithelial carcinoma (SEIC).
* Women older than 18 years of age.
* Women with understanding of Dutch or English language in reading and writing.

Exclusion Criteria:

* Diagnosis with a different type of endometrial neoplasm or invasive carcinoma.
* Previous and/or current treatment for another malignancy (<2 year before diagnosis of SEIC).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals with an uterus and endometrial disease are eligible.
Study Population: Women with serous endometrial intra-epithelial carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2035-04-01 (Estimated); Study Completion 2035-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5 years
  Survival without recurrence of endometrial neoplasm

SECONDARY OUTCOMES:
Overall survival | 5 years
Health-related quality of life | 5 years
  Assessed through EORTC questionnaires Assessed through three different questionnaires: EORTC-QLQ-C30 + QLQ-EN24 (together a total of 54 multiple-choice questions with a scale of 1-4 of severity of complaints) and EQ-5D-5L (multiple-choice, scale of severity, all different items will be entered in the digital database)
Adverse events | 5 years
  Any adverse event related to the treatment of SEIC

CONTACTS AND LOCATIONS:
Overall Officials: Heleen J. van Beekhuizen, Principal Investigator — Erasmus Medical Center, Cancer Institute
Locations (1):
- Franciscus Gasthuis & Vlietland, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slaager C, Hofhuis W, Hoogduin KJ, Ewing-Graham PC, van Beekhuizen HJ. Serous endometrial intra-epithelial carcinoma: an observational study. Int J Gynecol Cancer. 2023 Jun 5;33(6):905-914. doi: 10.1136/ijgc-2023-004281. PMID 37130624